CLINICAL TRIAL: NCT01785888
Title: A Diagnostic Study of European and Japanese Advanced NSCLC Patients to Evaluate Suitable Sample Types for EGFR Testing,
Brief Title: Europe-Japan Diagnostic Study for EGFR Testing
Acronym: ASSESS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7913C00070
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: EGFR Mutation Status in aNSCLC Patients (Locally Advanced and/or Metastatic Disease) With Adenocarcinoma and Non-adenocarcinoma Histologies.
Keywords: EGFR,; aNSCLC,; mutation status,; diagnostic study,; Europe,; Japan
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour samples (biopsy or citology) Blood (plasma) samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Locally advanced/metastatic NSCLC pts.: Patients(pts.) with locally advanced (stage IIIA/B) or metastatic NSCLC who have not received any local or systemic chemotherapy, and are not eligible for curative treatment (including surgery and chemoradiotherapy)

SUMMARY:
This is a non-interventional diagnostic, international, multicenter and non-comparative study of EGFR mutation status in aNSCLC patients (locally advanced and/or metastatic disease) with adenocarcinoma and non-adenocarcinoma histologies. This study will be conducted in Japan and Europe and will assess the concordance of EGFR mutation status derived from tumour samples and blood based circulating free DNA. The data generated will inform the use of less-invasive sample types in diagnostic practice. The study also aims to assess the current status of EGFR mutation testing across Japan and Europe and gaps in currently available data including EGFR mutation frequency in particular populations and demographic subgroups, EGFR mutation frequency in histological subtypes of NSCLC, EGFR mutation test process and methodology, utility of multiple sample types in the assessment of EGFR mutation status, and impact of EGFR mutation status on therapy choice. The data may be used to drive improvements to the EGFR mutation testing process, ensuring that patients have access to testing and are treated appropriately on the basis of the molecular features of their disease.

DETAILED DESCRIPTION:
A diagnostic Study of European and Japanese advanced NSCLC patients to evaluate suitable sample types for EGFR testing,

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older in Europe and aged 20 years and older in Japan
* Histological or cytological confirmed locally advanced NSCLC (stage IIIA/B) not suitable for curative treatment or metastatic (stage IV) NSCLC.
* Newly diagnosed patients with locally advanced and/or metastatic NSCLC who are systemic treatment Naïve (i.e. no chemotherapy or EGFR-TKI) or patients with recurrent disease who have previously received adjuvant chemotherapy (not including EGFR-TKI)
* Provision of diagnostic cancer tissue or cytology sample upon inclusion
* Provision of a routine blood sample

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease
* Evidence of any other significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study
* Pregnancy or breast-feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with locally advanced (stage IIIA/B) or metastatic NSCLC who are newly diagnosed, have not received any local or systemic chemotherapy. Locally advanced patients should not be eligible for curative treatment (including surgery and chemoradiotherapy).
  * Patients who have newly diagnosed locally advanced (stage IIIA/B) NSCLC who are not eligible for curative treatment (including surgery and chemoradiotherapy) or metastatic NSCLC and have not received systemic chemotherapy. Previous or planned palliative radiotherapy is allowed.
  * Patients who have had surgical resection with or without adjuvant chemotherapy and have experienced recurrent disease.
Sampling Method: Probability Sample
Enrollment: 1311 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Determination of the level of concordance between EGFR mutation status obtained via tissue/cytology and blood (plasma) based testing. | From randomization until study completion, assessed up to 17 months

SECONDARY OUTCOMES:
Determination of the EGFR mutation frequency (including mutation subtypes) in patients with advanced NSCLC (aNSCLC) of adenocarcinoma and non-adenocarcinoma histologies. | From randomization until study completion, assessed up to 17 months.
Describe the first line therapy choice following EGFR mutation testing. | From randomization until study completion, assessed up to 17 months.
Describe the second line therapy choice following discontinuation of first line treatment for patients confirmed as EGFR mutation positive via tissue/cytology. | From randomization until study completion, assessed up to 17 months.
Summary of EGFR mutation testing practices in terms of methods, sample types, success rate, mutation detection rate, testing turnaround time and reasons for not testing. | From randomization until study completion, assessed up to 17 months.
Determination of the correlation between EGFR mutation status from tumour and demographic data and disease status. | From randomization until study completion, assessed up to 17 months.
Determination of the correlation between EGFR mutation status derived from plasma (blood) and demographic data and disease status. | From randomization until study completion, assessed up to 17 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rose McCormack, PhD, Study Director — AstraZeneca
Locations (57):
- France (9):
  - Research Site, Compiègne
  - Research Site, Gap
  - Research Site, Le Mans
  - Research Site, Longjumeau
  - Research Site, Meaux
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Michel
  - Research Site, Saint-Quentin
  - Research Site, Villefranche-sur-Saône
- Germany (10):
  - Research Site, Buch
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hemer
  - Research Site, Karlsruhe
  - Research Site, Löwenstein
  - Research Site, Münnerstadt
  - Research Site, Nuremberg
  - Research Site, Solingen
- Italy (8):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Lecce
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Orbassano (TO)
  - Research Site, Perugia
  - Research Site, Rome
- Japan (8):
  - Research Site, Hirakata
  - Research Site, Iizuka
  - Research Site, Kanazawa
  - Research Site, Mibu
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Tokyo
  - Research Site, Toyonaka
- Netherlands (6):
  - Research Site, 's-Hertogenbosch
  - Research Site, Arnhem
  - Research Site, Bergen op Zoom
  - Research Site, Breda
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Cruces
  - Research Site, Donostia / San Sebastian
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Pontevedra
- Sweden (3):
  - Research Site, Gävle
  - Research Site, Karlstad
  - Research Site, Uppsala
- United Kingdom (6):
  - Research Site, Cardiff
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sheffield

REFERENCES:
- See also: CSR_Synopsis_D7913C00070.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=597&filename=CSR_Synopsis_D7913C00070.pdf
- See also: redacted protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=597&filename=ASSESS_redacted_protocol.pdf